CLINICAL TRIAL: NCT04831099
Title: Testosterone Treatment in a Patient With 17β-hydroxysteroid Dehydrogenase Type 3 Deficiency: an N-of-1 Study
Acronym: N-of-1 DSD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, dr. Laura C. G. de Graaff-Herder, Principal investigator, Erasmus Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N-of-1 DSD
Record Dates: First submitted 2021-03-26; First posted 2021-04-05 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-04

CONDITIONS: Disorder of Sex Development, 46,XY
Keywords: 17-beta-hydroxysteroid dehydrogenase type 3 deficiency
MeSH Terms: conditions — Disorder of Sex Development, 46,XY | interventions — Testosterone

STUDY DESIGN:
Intervention Model Description: N-of-1 study: cross-over study in 1 patient with 2 cycles that each consists of 2 periods (one period of placebo and one period of active treatment).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The participant and investigator are blinded. The investigator is also the care provider and investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Testosterone (Experimental): Testosterone gel (20 mg/day) for 8 weeks per period.
  Interventions: Drug: Testosterone gel
- Placebo (Placebo Comparator): Placebo gel (20 mg/day) for 8 weeks per period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Testosterone gel — The route of administration is transdermal.
  Other Names: AndroGel
  Arms: Testosterone
Drug: Placebo — The route of administration is transdermal
  Arms: Placebo

SUMMARY:
A 38-year old women with a 46,XY disorder of sex development (DSD) based on a 17β-hydroxysteroid dehydrogenase type 3 deficiency (17β-HSD3) was seen at the department of Internal Medicine-Endocrinology at the Erasmus MC, Rotterdam, the Netherlands.

The patient presented with fatigue, concentration problems and feelings of restlessness. In the past, the patient had undergone a gonadectomy at 9 months of age. In a follow-up visit at the outpatient clinic, the patient mentioned that friends with DSD had successfully been treated with testosterone and the patient requested testosterone treatment for her complaints.

In the literature, nothing is known about the usefulness of testosterone treatment for women with 17β-HSD3. For other forms of 46,XY DSD like complete androgen insensitivity syndrome (CAIS), limited data are available about testosterone treatment. Two studies have compared the effects of estrogen and testosterone replacement therapy on psychological wellbeing, quality of life (QoL) and sexual function in women with CAIS. The results were not conclusive, as one of them found a positive effect of testosterone replacement therapy on sexual function compared to estrogen, whereas the other study found no differences.

In order to evaluate the effect of testosterone treatment independent of a possible placebo effect, the usefulness of testosterone treatment in this individual patient with 17β-HSD3 will be investigated in an N-of-1 trial in order to improve the clinical care for this patient.

The primary objective is to determine the efficacy of testosterone treatment for fatigue on an individual level in a patient with 17β-HSD3 as assessed with the Checklist Individual Strength (CIS-20).

DETAILED DESCRIPTION:
A 38-year old women with a 46,XY disorder of sex development (DSD) based on a 17β-hydroxysteroid dehydrogenase type 3 deficiency (17β-HSD3) was seen at the department of Internal Medicine-Endocrinology at the Erasmus MC, Rotterdam, the Netherlands.

17β-HSD3 is a rare disorder characterized by a (despite the presence of a Y chromosome) female habitus in almost all newborns, with congenital agenesis of the uterus and ovaries. During puberty, patients with 17β-HSD3 often develop secondary male characteristics, such as deepening of the voice, male pattern body hair, and clitoromegaly.

The patient presented with fatigue, concentration problems and feelings of restlessness. In the past, the patient had undergone a gonadectomy at 9 months of age. In a follow-up visit at the outpatient clinic, the patient mentioned that friends with DSD had successfully been treated with testosterone and the patient requested testosterone treatment for her complaints. The patient was aware of the fact that the positive effect noticed by the patients' friends could be (partly) explained by placebo effect.

In the literature, nothing is known about the usefulness of testosterone treatment for women with 17β-HSD3. For other forms of 46,XY DSD like complete androgen insensitivity syndrome (CAIS), limited data are available about testosterone treatment. Two studies have compared the effects of estrogen and testosterone replacement therapy on psychological wellbeing, quality of life (QoL) and sexual function in women with CAIS. The results were not conclusive, as one of them found a positive effect of testosterone replacement therapy on sexual function compared to estrogen, whereas the other study found no differences.

In order to evaluate the effect of testosterone treatment independent of a possible placebo effect, the usefulness of testosterone treatment in this individual patient with 17β-HSD3 will be investigated in an N-of-1 trial in order to improve the clinical care for this patient.

The primary objective is to determine the efficacy of testosterone treatment for fatigue on an individual level in a patient with 17β-HSD3 as assessed with the Checklist Individual Strength (CIS-20).

Secondary objectives are to determine the effect of testosterone treatment on the QoL (5-level EQ-5D), testosterone, dehydroepiandorosterone (DHEA), and estradiol levels, on bone density, and on specific personalized goals that are important to the patient and her environment (Goal Attainment Scaling). To monitor the safety of testosterone treatment, hematocrit levels will be measured and the occurrence of adverse events will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

- N/A

Exclusion Criteria:

- N/A

The study is especially designed for a specific female patient. The patient is 38 years old at the moment. Since the study is especially designed for this patient, there are no formal inclusion and exclusion criteria.

Min Age: 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2022-07-26 (Estimated); Study Completion 2022-07-26 (Estimated)

PRIMARY OUTCOMES:
Fatigue (Checklist of Individual Strength) | Baseline to 420 days
  Fatigue is measured with the Checklist of Individual Strength (CIS-20). The CIS-20 consists of 20 questions. The score ranges from 20 - 140. A score of 27-35 means increased fatigue. A score >35 means extreme fatigue.

SECONDARY OUTCOMES:
Quality of Life (5-level EQ-5D) | Baseline to 420 days
  Quality of life is measured with the 5-level EQ-5D (EQ-5D-L5). The range of the EQ-5D-5L is from 0 to 100. A higher score means a better outcome.
Laboratory levels | Baseline to 420 days
  The following laboratory levels will be measured:
  * Testosterone (nmol/L)
  * Dehydroepiandorosterone (DHEA) (micromol/L)
  * Estradiol (pg/mL)
  * Hematocrit (%)
Bone density | Baseline to 420 days
  Dual Energy X-ray Absorptiometry scan will be performed to measure bone density.
Goal attainment scaling | Baseline to 420 days
  GAS is an individualized outcome measure in which several personal goals and the corresponding scaling are defined in consultation with the patient. The scaling is standardized, which makes it possible to reliably measure the change in the situation of the patient. The levels range from -3 to +2. A higher level means a better outcome. The predefined personal goals are a measure of the effectivity of the treatment. If possible, three goals will be set.
Number of adverse events | Baseline to 450 days
  All adverse events that occur from start of treatment until 30 days after last administration will be described to assess the safety of testosterone treatment. Adverse events are defined as any undesirable experience occurring during the study, whether or not considered related to testosterone treatment

CONTACTS AND LOCATIONS:
Overall Officials: Laura de Graaff, MD, PhD, Principal Investigator — Department of Internal Medicine - Endocrinology, Erasmus MC, Rotterdam, the Netherlands
Locations (1):
- Erasmus MC, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data is available upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: The data will become available after completion of the study and only upon reasonable request and with permission of the participant.
Access Criteria: A motivated request.